CLINICAL TRIAL: NCT05559359
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 3 Study to Assess the Efficacy, Safety and Pharmacokinetics of Lebrikizumab Compared to Placebo in Participants 6 Months to <18 Years of Age With Moderate-to-Severe Atopic Dermatitis
Brief Title: A Study of Lebrikizumab (LY3650150) in Participants 6 Months to <18 Years of Age With Moderate-to-Severe Atopic Dermatitis
Acronym: ADorable-1
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Dermira, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18265; J2T-MC-KGBI (Other: Eli Lilly and Company); DRM06-AD13 (Other: Dermira Inc); 2021-005232-29 (EudraCT Number); 2022-501476-25-00 (Other: EU Trial Number)
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Atopic Dermatitis; Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — lebrikizumab; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Lebrikizumab (Cohort 1) (Experimental): Participants who are 6 years to <18 years of age, 12 years to <18 years of age who weigh <40 kilogram (kg) or 6 years to <12 years of age (may weigh ≥40 kg) will receive a loading dose and then subsequent doses by subcutaneous (SC) injections with a topical corticosteroid (TCS).
  Dosing will be based on weight.
  Interventions: Drug: Lebrikizumab; Drug: Topical Corticosteroid (TCS)
- Lebrikizumab (Cohort 2) (Experimental): Participants who are 6 months to <6 years of age, 2 years to <6 years of age or 6 months to <2 years of age will receive a loading dose of lebrikizumab and then subsequent doses by SC injections with a TCS.
  Dosing will be based on weight.
  Interventions: Drug: Lebrikizumab; Drug: Topical Corticosteroid (TCS)
- Placebo (Placebo Comparator): Participants will receive placebo matching lebrikizumab by SC injections with a TCS.
  Interventions: Drug: Placebo; Drug: Topical Corticosteroid (TCS)

INTERVENTIONS:
Drug: Lebrikizumab — Administered SC
  Other Names: LY3650150; DRM06
  Arms: Lebrikizumab (Cohort 1); Lebrikizumab (Cohort 2)
Drug: Placebo — Placebo given SC
  Arms: Placebo
Drug: Topical Corticosteroid (TCS) — TCS administered

SUMMARY:
The main purpose of this study is to measure the effect, safety and how well the body absorbs lebrikizumab in pediatric participants 6 months to <18 years of age with moderate-to-severe atopic dermatitis (AD).

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of AD prior to screening as stated in the criteria by the American Academy of Dermatology for at least,

  * 12 months if participants are ≥6 years of age
  * 6 months if participants are 2 to <6 years of age
  * 3 months if participants are 6 months to <2 years of age.
* Have an EASI score ≥16 at the screening and baseline
* Have an IGA score ≥3 (scale of 0 to 4) at the screening and baseline
* Have ≥10% BSA of AD involvement at the screening and baseline.

Exclusion Criteria:

* Are currently enrolled or have participated within the last 8 weeks in a clinical study involving an investigational intervention or any other type of medical research judged not to be scientifically or medically compatible with this study.
* Treatment with the following prior to the baseline:
* An investigational drug within 8 weeks or less than 5 half-lives, whichever is longer.
* Dupilumab within 8 weeks. Note: The enrollment of participants with prior use of Dupilumab will be limited to <20%.
* Treatment with a topical investigational drug within 2 weeks prior to the baseline.
* Have received a Bacillus Calmette-Guerin vaccination or treatment within less than 4 weeks before randomization.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 367 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2026-01-14 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with an Investigator Global Assessment (IGA) score 0 or 1 and a Reduction ≥2 points from Baseline | Baseline to Week 16
  EASI-75 is a co-primary endpoint with IGA.
Percentage of Participants Achieving Eczema Area and Severity Index-75 (EASI-75) ≥75% Reduction from Baseline in EASI Score | Baseline to Week 16
  IGA is a co-primary endpoint with EASI-75.

SECONDARY OUTCOMES:
Percentage of Participants Achieving EASI-90, a ≥90% Reduction from Baseline in EASI Score | Baseline to Week 16
Percentage of Participants with a Pruritus Numeric Rating Score (NRS) of ≥4 points at Baseline Who Achieve a ≥4-point Reduction from Baseline | Baseline to Week 16
Percentage of Participants with a cDLQI of ≥6 points at Baseline Achieving ≥6-point Improvement in cDLQI from Baseline to Week 16 | Baseline to Week 16
Percentage Change from Baseline in EASI Score | Baseline, Week 16
Percentage Change from Baseline in Pruritus NRS Score | Baseline, Week 16
Change from Baseline in Children Dermatology Life Quality Index (cDLQI) | Baseline, Week 16
Mean Change from Baseline in Worst Scratch/Itch Numeric Rating Score (WSI-NRS) | Baseline, Week 16
Change from Baseline in Body Surface Area (BSA) | Baseline, Week 16
Percentage Change from Baseline in Scoring Atopic Dermatitis (SCORAD) | Baseline, Week 16
Percentage of Participants Achieving EASI-50, a ≥50% Reduction from Baseline in EASI Score | Baseline to Week 16
Pharmacokinetics (PK): Average Serum Lebrikizumab Concentration | Week 14
Percentage of Participants with Positive Responses by the Modified Subcutaneous Administration Assessment Questionnaire (mSQAAQ) | Week 14
Percentage of Participants with a Worst Scratching/Itching NRS of ≥4 points at Baseline Who Achieve a ≥4-point Reduction from Baseline to Week 16 | Baseline to Week 16
Change from Baseline in SCORAD | Baseline, Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (85):
- United States (21):
  - Clinical Research Center of Alabama, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Research Trials, North Little Rock, Arkansas
  - First OC Dermatology, Fountain Valley, California
  - Antelope Valley Clinical Trials, Lancaster, California
  - Dermatology Research Associates, Los Angeles, California
  - Integrative Skin Science and Research, Sacramento, California
  - Rady's Children Hospital San Diego - Dermatology, San Diego, California
  - UConn Health, Farmington, Connecticut
  - Solutions Through Advanced Research, Jacksonville, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Treasure Valley Medical Research, Boise, Idaho
  - Northwestern University, Chicago, Illinois
  - Allergy & Asthma Specialists, P.S.C., Owensboro, Kentucky
  - Respiratory Medicine Research Institute of Michigan, PLC, Ypsilanti, Michigan
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Psoriasis Treatment Center of Central New Jersey, East Windsor, New Jersey
  - Dermatologists of Central States, LLC, Fairborn, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Argentina (6):
  - CONEXA Investigacion Clinica S.A., Buenos Aires
  - Instituto de Neumonología Y Dermatología, Buenos Aires
  - Derma Internacional, Buenos Aires
  - Psoriahue, Buenos Aires
  - Fundación Respirar, Buenos Aires
  - Fundacion Estudios Clinicos, Rosario
- Australia (4):
  - Cornerstone Dermatology, Coorparoo
  - Sydney Children's Hospital, Randwick
  - The Children's Hospital at Westmead, Westmead
  - Veracity Clinical Research, Woolloongabba
- Brazil (7):
  - Fundação Pio XII - Hospital de Câncer de Barretos, Barretos
  - Centro de Pesquisa Sao Lucas, Campinas
  - Hospital de Clinicas de Porto Alegre, Porto Alegre
  - Hospital de Clínicas de Ribeirão Preto, Ribeirão Preto
  - IBPClin - Instituto Brasil de Pesquisa Clínica, Rio de Janeiro
  - Faculdade de Medicina do ABC, Santo André
  - Clinica de Alergia Martti Antila, Sorocaba
- Canada (2):
  - Dermatology Research Institute, Calgary
  - DermEdge Research, Mississauga
- Fakultni nemocnice Bulovka, Prague, Czechia
- Germany (5):
  - Fachklinik Bad Bentheim, Bad Bentheim
  - Rosenpark Research GmbH, Darmstadt
  - Universitaetsklinikum Carl Gustav Carus Dresden, Dresden
  - Universitätsklinikum Frankfurt, Frankfurt
  - Universitätsklinikum Münster, Münster
- Japan (12):
  - Asahikawa Medical University Hospital, Asahikawa
  - Fukuyama City Hospital, Fukuyama
  - Osaka Habikino Medical Center, Habikino
  - Hiroshima University Hospital, Hiroshima
  - Ina Central Hospital, Ina
  - Enomoto Clinic, Kumagaya
  - University Hospital,Kyoto Prefectural University of Medicine, Kyoto
  - Okayama City General Medical Center Okayama City Hospital, Okayama
  - National Hospital Organization Sagamihara National Hospital, Sagamihara
  - Dermatology and Ophthalmology Kume Clinic, Sakai
  - Sugamo Sengoku Dermatology, Toshima City
  - Fujita Health University, Toyoake
- Mexico (9):
  - Scientia Investigacion Clinica S.C., Chihuahua City
  - PanAmerican Clinical Research - Cuernavaca, Cuernavaca
  - Hospital de Jesús Nazareno, Mexico City
  - Trials in Medicine, Mexico City
  - Hospital Infantil de Mexico Federico Gomez, Mexico City
  - Eukarya PharmaSite, Monterrey
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey
  - Arké SMO S.A de C.V, Veracruz
  - Instituto Dermatologico de Jalisco, Zapopan
- Poland (4):
  - Centrum Badan Klinicznych PI-House sp. z o.o., Gdansk
  - Diamond Clinic, Krakow
  - "DERMED" Centrum Medyczne Sp. z o.o., Lodz
  - Centrum Medyczne Evimed, Warsaw
- Spain (7):
  - Hospital Sant Joan de Déu, Esplugues de Llobregat
  - Hospital Universitario de Gran Canaria Doctor Negrín, Las
  - Grupo Pedro Jaén, Madrid
  - Hospital Infantil Universitario Niño Jesús, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Clinica Universidad de Navarra, Pamplona
- Taiwan (7):
  - National Taiwan University Hospital - Hsinchu branch, Hsinchu
  - Chang Gung Memorial Hospital at Kaohsiung, Kaohsiung Niao Sung Dist
  - Chung Shan Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital-Taipei, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: A Study of Lebrikizumab (LY3650150) in Participants 6 Months to <18 Years of Age With Moderate-to-Severe Atopic Dermatitis — https://trials.lilly.com/en-US/trial/362456